CLINICAL TRIAL: NCT04304690
Title: COVID-19 Seroconversion Among Medical and Paramedical Staff in Emergency, ICU and Infectious Disease Services During the 2020 Epidemic
Brief Title: COVID-19 Seroconversion Among Front Line Medical and Paramedical Staff in Emergency, Intensive Care Units and Infectious Disease Departments During the 2020 Epidemic
Acronym: SEROCOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP200310
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Sars-CoV2
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- caregiver (Other): caregivers from emergency, ICU, virology and infectious disease services
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample — 2 blood samples at T0 and 3 months

SUMMARY:
The epidemic due to the Sars-CoV2 virus is spreading in France, without knowning precisely since when the virus has actually circulated on the territory. Data from China but also systematic samples taken from the passengers of the Diamond Princess boat also report almost 50% of asymptomatic forms of Covid-19. The medical and paramedical staff of the front-line services for the care of patients infected with Covid-19 are in fact potentially exposed to the risk of occupational contamination due to the large number of patients treated, including in the pre-epidemic phase. Therefore, and despite the application of standard protective measures, it is possible that a certain number of these personnel already have or will contract Covid-19 disease, including in its asymptomatic form.

DETAILED DESCRIPTION:
The epidemic due to Sars-CoV2 is spreading in France, without it being knowning precisely since when the virus actually circulated on the territory. Data from China but also systematic samples taken from the passengers of the boat Diamond Princess also report almost 50% of asymptomatic forms of Covid-19. Medical and paramedical staff are in fact potentially exposed to the risk of professional contamination, with probably a different risk between the first-line referent hospitals and the others, due to the large number of patients treated in the first, including in the pre-epidemic phase (average of 190 consultants per day at the emergency department Pitié-Salpêtrière for example). Therefore, and despite the application of standard protective measures, it is possible that a certain number of these personnel already have or will contract Covid-19 disease, including in its asymptomatic form. Knowledge of this seroconversion rate, if it is found to be higher than that of the general population, could lead to a review of the measures to protect personnel from other emerging infectious risks.

ELIGIBILITY:
Inclusion Criteria:

* Any permanent medical or paramedic staff of participating services who have given written consent to participate
* Having a social security insurance.

Exclusion Criteria:

* Non-permanent staff (occasional staffing), administrative staff, technical staff of participating services.
* Staff who were not active during the inclusion period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1177 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Quantify the proportion of patients with documented Sars-CoV2 infection among medical and paramedical staff | 3 months
  Sars-CoV2 seroconversion is defined by a T0 sample with no specific antibody (negative) and M3 sample with the presence of specific IgG.

SECONDARY OUTCOMES:
Identification of risk factors for seroconversion | 3 months
  "Age, gender, type of staff, medical staff: resident, Clinic Chief or University Hospital Assistant (CCA / AHU), Associate Practitioner (PA), Contractual Hospital Practitioner (PHC), Hospital Practitioner (PH), Lecturer-Hospital Practitioner (MCU-PH) , University Professor-Hospital Practitioner (PUPH) non-medical staff: nursing assistants (AS), nurses (IDE), physiotherapist, managers, others, Seniority in the profession (number of years) Service tenure (years), Night, day, day or mixed work, Type of service: emergency department, infectious disease service, ICU), Type of hospital (firstline reference hospital or not), Documented contact with a confirmed patient."
Quantify the proportion of asymptomatic infections among staff who have seroconverted | 3 months
  "Seroconversion without clinical manifestation (fever, body aches, headache, sweating, chills + respiratory symptoms (cough dyspnea, sputum) or digestive (nausea / vomiting diarrhea abdominal pain) reported via the weekly self-monitoring booklet.
  The asymptomatic characteristics will be determined by an adjudication committee, in the light of the weekly self-monitoring notebooks, without knowing the results of the serologies."
" Describe symptomatic infections for personnel developing acute clinical (respiratory or digestive) viral syndrome " | 3 months
  "Description of symptomatic infections
  * Clinical manifestations associated with seroconversion.
  * On the intermediate sample if necessary, performed within 10 days of the start of a clinical picture compatible with an acute Sars-CoV2 infection (fever, body aches, headache, sweating, chills + respiratory picture (cough dyspnea, sputum, ) or digestive (nausea / vomiting diarrhea abdominal pain) "

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Pitié Salpetrière, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hausfater P, Boutolleau D, Lacombe K, Beurton A, Dumont M, Constantin JM, Ghosn J, Combes A, Cury N, Guedj R, Djibre M, Bompard R, Mazerand S, Pourcher V, Gimeno L, Marois C, Teyssou E, Marcelin AG, Hajage D, Tubach F. Cumulative incidence of SARS-CoV-2 infection and associated risk factors among frontline health care workers in Paris: the SEROCOV cohort study. Sci Rep. 2022 May 4;12(1):7211. doi: 10.1038/s41598-022-10945-y. PMID 35508515